CLINICAL TRIAL: NCT03699072
Title: A Multi-centre, Pilot, Prospective Trial of DermaRep™ Device in the Treatment of Venous Leg Ulcers
Brief Title: DermaRep™ Device in the Treatment of Venous Leg Ulcers
Acronym: DermaRep™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biovotec AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BV-CP-01
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: DermaRep™ Wound Contact Device — Treatment of venous leg ulcers once weekly for 8 weeks along with standard of care dressings

SUMMARY:
This is a First in Human clinical study on the safety and effectiveness of DermaRep™ wound contact dressing. Patients with venous leg ulcers will be treated with standard of care dressings and compression for 4 weeks to establish a baseline wound healing response. All patients will then be treated with DermaRep™ wound contact dressing in addition to standard of care for a further 8 weeks. If the wound has not healed, patients will continue treatment with standard of care only for a further 4 weeks. All patients will be assessed at the 16 week timepoint, the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18 years of age
* The patient is male and female not pregnant or lactating and using contraception
* The patient has a confirmed venous leg ulcer with:Confirmed actively managed reflux; No exposed tendon or bone; Ulcer surface area between 2cm2 and 80cm; ABPI>0.8
* The patient agrees to abstain from enrolment in any other clinical trial for the duration of the study
* The patient is able to understand the aims and objectives of the trial and is willing to consent

Exclusion Criteria:

* Study treatment area has exposed bone or tendon
* Poorly controlled diabetes
* Arterial insufficiency (ABPI<0.8)
* Pregnant/lactating females (tested as per institutional requirements)
* The patient has a severe dermatological disorder (e.g. severe psoriasis, epidermolysis bullosa, pyoderma granulosum)
* The patient is unable to follow the procedures set by the protocol
* The patient has a history of any significant cardiac, pulmonary, renal. hepatic, neurological and/or immune dysfunction that in the opinion of the investigator may compromise patient safety or study objectives
* The patient is taking any known medications that in the opinion of the investigator may compromise patient safety or the study objectives
* The patient has any known allergies to any of the device materials to be used in the trial (egg allergy)
* The patient is a vulnerable or protected adult
* The patient is unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events following DermaRep™ treatment | 12 weeks
  Potential adverse events following DermaRep™ treatment will be compared to the pre-treatment phase, the 4 week run-in period. Adverse events will include active bleeding, clinical infection and device deficiencies.

SECONDARY OUTCOMES:
Evaluation of the performance of DermaRep™ in rate of wound healing. | 12 weeks
  Qualitative evaluation of wound healing progression will be assessed visually by the treating clinician
Assessment of Wound Pain | 12 weeks
  Wound pain will be assessed using a VAS score.
DermaRep™ Dressing Application | 12 weeks
  Pain on dressing changes will be assessed using a VAS score
Wound coverage | 12 weeks
  Wound coverage will be calculated as a percentage from baseline to the end of the study using wound grids for area measurement
Comparison of healing between the run-in period and the treatment period | 12 weeks
  The rate of progression in wound healing during the treatment phase relative to the pre-treatment run-in phase will be assessed by surface area measurement using wound grids.
Wounds healed at 12 weeks | 12 weeks
  The number of wounds healed at the final assessment will be assessed.
Reduction in wound area/volume | 12 weeks
  The % reduction in area and volume of the wound will be assessed by measurement with wound grids and a ruler.
Time to healing | 12 weeks
  Time to healing for healed wounds will be assessed in weeks.
Exudate levels | 12 weeks
  Exudate levels will be assessed qualitatively (low, medium, high) by the treating clinician.
Condition of the surrounding skin | 12 weeks
  The condition of the surrounding skin will be described qualitatively by the treating clinician

CONTACTS AND LOCATIONS:
Overall Officials: Kevin G Mercer, MD, Principal Investigator — Bradford Teaching Hospitals NHS Foundation Trust
Locations (6):
- United Kingdom (6):
  - Bradford Royal Infirmary, Bradford
  - Countess of Chester Hospital, Chester
  - Royal Free Hospital, London
  - Imperial College Charing Cross Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Northern General Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided